CLINICAL TRIAL: NCT03569930
Title: Irritation and Anal Bleeding in Patients Affected by Hemorrhoids: Comparative Evaluation of Three Different Treatments.
Brief Title: Irritation and Anal Bleeding in Patients Affected by Hemorrhoids.
Acronym: IR-AN-BLEED
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Massimo Chiaretti, Clinical Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URomLS-5
Record Dates: First submitted 2018-05-08; First posted 2018-06-26 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-05

CONDITIONS: Hemorrhoids
Keywords: Flavonoid-based supplements; Centella asiatica; Hemorrhoids; defecation; bleeding; pain
MeSH Terms: conditions — Hemorrhoids; Hemorrhage; Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard (Experimental): standard of care (diet rich in water and vegetable fibers, hygienic)
  Interventions: Behavioral: standard of care
- ProtFlav (Experimental): oral supplements (flavonoid-based supplements - ProtFlav) will be added to standard of care
  Interventions: Drug: flavonoid-based supplements
- ProtCent (Experimental): anal application of a Centella based cream (Centella asiatica - ProtCent) will be added to standard of care
  Interventions: Drug: Centella Complex

INTERVENTIONS:
Drug: flavonoid-based supplements — Ingredients: soybean oil (glycine max), edible gelatin, rutin, borage seed oil (borago officinalis), pineapple dry extract (ananas sativus), glycerol, thickeners (mono and diglycerides of fatty acids), emulsifier (soy lecithin).
  Arms: ProtFlav
Drug: Centella Complex — The components are: Centella Asiatica, Beta-glucan, Arnica, Aloe Vera, Menthol, Devil's claw, perform actions useful to alleviate the painful symptomatology, restore the tone of the venous wall, assist the treatment of microcirculatory damage.
  Arms: ProtCent
Behavioral: standard of care — diet rich in water and vegetable fibers, hygienic and anal dilator
  Arms: Standard

SUMMARY:
Haemorrhoidal disease is an increasingly frequent benign condition, able to negatively affect the quality of working and relationship life in affected individuals.The primary objective of the study is the comparative assessment of the time necessary for the disappearance of bleeding comparatively in the three different therapies (controls, ProtFlav and ProtCent) to identify, if any, the most effective treatment, in terms of time reduction for the disappearance of bleeding in subjects affected by haemorrhoidal disease.

Patients enrolled will be randomized into 3 groups:

1. the control group in which the patients will be subjected to the standard therapeutic care (diet rich in water and vegetable fibers, hygienic),
2. interventional group "ProtFlav": in which oral supplements (flavonoid-based supplements - ProtFlav) will be added to standard of care
3. interventional group "ProtCent": in which an anal application of a Centella based cream (Centella asiatica - ProtCent) will be added to standard of care

DETAILED DESCRIPTION:
Haemorrhoidal disease is an increasingly frequent benign condition, able to negatively affect the quality of working and relationship life in affected individuals.The primary objective of the study is the comparative assessment of the time necessary for the disappearance of bleeding comparatively in the three different therapies (controls, ProtFlav and ProtCent) to identify, if any, the most effective treatment, in terms of time reduction for the disappearance of bleeding in subjects affected by haemorrhoidal disease.

Secondary objectives are the evaluation of the longitudinal trend in time of anal irritation measured with the VAS scale and the study of the longitudinal performance of BMI (Body Mass Index).

The patients enrolled in the protocol will be randomized into 3 groups: the control group in which the patients will be subjected to a diet rich in water and vegetable fibers, hygienic care and anal dilator according to the traditional standardized scheme. The two experimental groups will be subjected to the same standard therapeutic scheme (diet rich in water and vegetable fibers, hygienic) of the controls, in addition to which will be added to oral supplements (group "ProtFlav") and local application as an anal cream (group "ProtCent"). Of the patients in the interventional groups, half will take flavonoid-based supplements (ProtFlav) and the other half will take supplements and anal cream based on Centella asiatica (ProtCent), as better specified below. All patients will be followed for a period of 8 weeks or otherwise until recovery (disappearance of irritation and stop bleeding).

ELIGIBILITY:
Inclusion Criteria:

* Male and female affected by acute haemorrhoidal disease
* Collaborating patients, able to understand

Exclusion Criteria:

* Women who are pregnant or have been breastfeeding;
* Previous colorectal surgery;
* Anal stenosis;
* Treatment (topical or systemic) with decongestants, diuretics, steroidal anti-inflammatory drugs or NSAIDs, antipyretics, antibiotics or antivirals for other reasons;
* Psychiatric and / or toxic employees;
* Age in completed years, less than 18 and over 85;
* If the patient's personal clinical record does not have at least two controls, it is excluded from the clinical study;
* Refusal to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
delta of time necessary for the disappearance of bleeding | 3 months
  comparative assessment of the time necessary for the disappearance of bleeding

SECONDARY OUTCOMES:
delta of Visual Analog Scale for Pain (VAS Pain) | 3 months
  longitudinal trend in time of anal irritation measured with the VAS scale for Pain (The VAS scale for pain is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (worst) to the right (best))
delta of BMI (Body Mass Index). | 3 months
  the longitudinal performance of BMI (Body Mass Index).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery "Paride Stefanini", University of Rome "La Sapienza", Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No